CLINICAL TRIAL: NCT01566045
Title: MRI/TRUS Fusion Guided Prostate Biopsy- An Improved Way to Detect and Quantify Prostate Cancer. A Phase III Study
Brief Title: MRI/TRUS Fusion Guided Prostate Biopsy- An Improved Way to Detect and Quantify Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02072012
Record Dates: First submitted 2012-02-22; First posted 2012-03-29 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core Needle TRUS biopsy (Transrectal ultrasound) (Active Comparator): Patient receiving core needle TRUS biopsy (Standard of care biopsy)
  Interventions: Procedure: Core Needle TRUS Needle biopsy (Transrectal ultrasound)
- Core Needle MRI/US fusion guided biopsy (Experimental): Patients receiving Standard of Care core needle TRUS biopsy will then receive the MRI / Ultrasound fusion core needle guided biopsy
  Interventions: Procedure: Core Needle MRI/US image fusion guided needle biopsy

INTERVENTIONS:
Procedure: Core Needle TRUS Needle biopsy (Transrectal ultrasound) — Standard of care 12-core TRUS sextant needle biopsy of the medial and lateral margins of the right and left apex, mid-gland and base of the prostate
  Other Names: Core Needle biopsy; TRUS needle biopsy (Transrectal ultrasound)
  Arms: Core Needle TRUS biopsy (Transrectal ultrasound)
Procedure: Core Needle MRI/US image fusion guided needle biopsy — Directed prostate needle biopsies at MR-image identified targets in addition to the standard ultrasound 12-14 core biopsies
  Other Names: Core Needle biopsy; MRI/US image fusion guided needle biopsy
  Arms: Core Needle MRI/US fusion guided biopsy

SUMMARY:
This study will determine if targeted (Magnetic Resonance (MR) / Ultrasound (US) fusion biopsy) plus conventional biopsy is superior to conventional biopsy alone in diagnosing subjects with prostate cancer.

DETAILED DESCRIPTION:
The efficacy of targeting lesions for surgery may be limited by the visibility of a target during the procedure. The successful outcome of surgical intervention depends upon accurate device placement, which may be very challenging in certain settings, such as when a kidney tumor only is visible for a brief moment during the transient arterial phase of a contrast injection, and soon disappearing on dynamic imaging.

Historically, prostate cancer was diagnosed by digitally guided trans-rectal prostate biopsies. With PSA (Prostate SPecific Antigen) screening and improvements in ultrasonography, trans-rectal ultrasound (TRUS) guided prostate biopsy have become the standard of care to screen and diagnose localized prostate cancer. Standard US 12-14 core prostate biopsy is now common practice, detecting cancer in 27% to 44% of patients.

Prostate MR imaging with the addition of an endorectal-coil probe and a 3 Tesla magnet dramatically improves diagnostic utility dramatically but biopsies are difficult, time-consuming, and require specialized equipment, which increases the cost significantly.

To meet this challenge TRUS images are overlaid on a previously obtained prostate MRI, combined with an electromagnetic tracking system. The urologist then performs directed prostate biopsies at MR-identified targets in addition to the standard 12-14 core biopsies.

This study will consist of comparison of the standard of care (TRUS guided prostate biopsy) with the protocol biopsy which consists of a TRUS guided prostate biopsy and a MR/US fusion tracked prostate biopsy. Each patient will act as their own control.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a pre-operative MRI performed in accordance with our NSHSLIJ/NIH MR prostate imaging guidelines.
2. Age greater than 18 years.
3. No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
4. The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.
5. Ability to tolerate conscious sedation (if procedure to be performed with conscious sedation, and without general anesthesia).
6. PSA > 2.5 or Abnormal digital rectal exam or current recommendations for biopsy from the American Urological Association
7. Pre-biopsy prostate MRI as described above, showing targetable lesions within 2 months of biopsy
8. Able to tolerate a TRUS guided biopsy

Exclusion Criteria:

1. Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study.
2. Patients unlikely able to hold reasonably still on a procedure table for the length of the procedure.
3. Inability to hold breath, if procedure will be performed with conscious sedation, and without general anesthesia.
4. Patients with pacemakers or automatic implantable cardiac defibrillators (contraindications to MRI)
5. Patients with uncorrectable coagulopathies.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Number of prostate lesions | Day 1
  To determine if the number of prostate lesions identified by targeted (MR / US fusion biopsy) plus conventional biopsy is statitically greater than the number of lesions identified conventional biopsy alone. The number of positive lesions identified by both techniques will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- The Arthur Smith Institute for Urology, New Hyde Park, New York, United States